CLINICAL TRIAL: NCT03636880
Title: Insomnia, Cognitive Impairment, and Decision Making Among Patients With Heart Failure:A Randomized Study of Brief Behavioral Treatment for Insomnia
Brief Title: Heart Failure Insomnia Treatment Study
Acronym: H-FITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Charles Emery PhD, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016H0451
Record Dates: First submitted 2018-08-08; First posted 2018-08-17 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Cardiac Failure; Congestive Heart Failure; Insomnia; Sleep Disorder; Sleep Initiation and Maintenance Disorders; Disorders of Initiating and Maintaining Sleep; Anxiety; Depression
Keywords: heart failure; insomnia; anxiety; depression; memory; attention; executive functioning; decision making; self-care; quality of life; functional status; walk test; sleep monitoring
MeSH Terms: conditions — Heart Failure; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Anxiety Disorders; Depression | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Baseline assessment is completed prior to randomization. Assessments conducted at 2 weeks and 6 months post-intervention are completed by an assessor blinded to participants' assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief treatment for insomnia (Experimental): Brief Behavioral Treatment for Insomnia (BBTI) is a manualized, individual intervention designed to modify sleep patterns to reduce insomnia and improve sleep quality and efficiency. Participants complete two in-person meetings and two booster telephone calls over a four-week period.
  Interventions: Behavioral: Brief treatment for Insomnia
- Sleep Monitoring (Active Comparator): Sleep Monitoring is an active comparator condition where participants track their sleep patterns for two weeks prior to the baseline and post-intervention assessments. They receive no contact from study staff during the intervening four-week period, except for a reminder call to begin completing the second sleep diary and to schedule the post-intervention assessment.
  Interventions: Behavioral: Sleep Monitoring

INTERVENTIONS:
Behavioral: Brief treatment for Insomnia — This behavioral intervention provides participants with an individualized plan to modify sleep patterns contributing to insomnia, as well as education about sleep hygiene and habits that help and hurt sleep.
  Other Names: BBTI
  Arms: Brief treatment for insomnia
Behavioral: Sleep Monitoring — This intervention involves using sleep diaries to track daily aspects of sleep, including bed time, wake time, hours of sleep, nighttime awakenings, daytime naps, and sleep quality.
  Arms: Sleep Monitoring

SUMMARY:
The purpose of this study is to compare a short, behavioral treatment for insomnia with sleep monitoring to determine whether these approaches are effective in reducing insomnia and improving sleep quality among patients with heart failure (HF). This study will also examine the relationship between insomnia and cognitive functioning in HF and the effects of the behavioral treatment on cognitive functioning, self-care, distress, HF symptoms, and functional status.

Participants will be randomly assigned to four-sessions of a behavioral treatment (Brief Behavioral Treatment for Insomnia; BBTI) or sleep monitoring.

DETAILED DESCRIPTION:
Comorbid insomnia is prevalent among heart failure (HF) patients and associated with poorer mental and physical functioning, including possible exacerbation of cognitive deficits. Initial investigations document the effectiveness of cognitive-behavioral therapy for the treatment of insomnia in HF. However, the high symptom burden of HF necessitates alternative interventions for these patients with fewer time and physical endurance demands.

Brief Behavioral Treatment for Insomnia (BBTI) is a four-session behavioral intervention that emphasizes stimulus control and sleep restriction techniques, along with providing education to patients about healthy sleep practices and behaviors that adversely affect sleep. The efficacy of BBTI has been previously documented in samples of older adults with insomnia, but the intervention has yet to be applied to a disease-specific patient population.

This study was designed to 1) evaluate the treatment effects of BBTI on insomnia among HF patients, 2) examine the relationship between insomnia, cognitive function, and decision-making in HF patients at baseline, and 3) evaluate the effects of BBTI on relevant correlates of insomnia in HF patients, including cognitive functioning, decision-making, distress, self-care, quality of life, and functional status.

Participants will be randomized to either the four-session behavioral intervention (BBTI) or a sleep monitoring condition. Measures of sleep (insomnia, sleep efficiency, sleep quality), cognitive functioning (memory, attention, executive functioning, and decision making), distress (anxiety and depression), HF-related quality of life, HF self-care, and functional status will be obtained from participants at baseline, post-intervention, and 6 months post-intervention. Repeated measures multivariate analysis of variance (MANOVA) will serve as the primary mode of data analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English
* Diagnosis of heart failure
* At least mild chronic insomnia

Exclusion Criteria:

* Restless legs syndrome
* Narcolepsy
* Perform night or rotating shift work
* Seizure disorder
* Excessive daytime sleepiness
* Current or past diagnosis of Bipolar disorder or psychotic disorder
* Significant cognitive impairments
* Untreated moderate to severe sleep apnea or high risk for sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | Change from pre-intervention to 2 weeks post-intervention
  Insomnia symptoms will be measured with the 7-item self-report Insomnia Severity Index (ISI). This measure assesses the severity of sleep-onset and sleep maintenance difficulties, sleep satisfaction, as well as associated daytime dysfunction and distress over the prior two weeks. Items are answered on a 5-point Likert-scale from 0 'not at all' to 4 'extremely'. Total scores range from 0 to 28, with higher scores reflective of greater insomnia severity. Scores of 8 or greater indicate the presence of at least mild clinical insomnia.
Sleep quality assessed by the PSQI | Change from pre-intervention to 2 weeks post-intervention
  Sleep quality will be measured with the 19-item self-report Pittsburgh Sleep Quality Index (PSQI). Seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction) are derived from the instrument which can then be summed to produce a total 'global' PSQI score ranging from 0 to 21. Total PSQI scores greater than 5 indicate poor sleep quality.
Sleep efficiency | Change from pre-intervention to 2 weeks post-intervention
  Sleep efficiency (SE) will be measured with two-week sleep diaries where participants log their daily bed and wake times, as well as the number of hours of sleep each night. SE will be calculated as the percentage of sleep time divided by time spent in bed, with higher percentages indicative of more efficient sleep.

SECONDARY OUTCOMES:
Insomnia severity | Pre-intervention
  Insomnia symptoms will be measured with the 7-item self-report Insomnia Severity Index (ISI). This measure assesses the severity of sleep-onset and sleep maintenance difficulties, sleep satisfaction, as well as associated daytime dysfunction and distress over the prior two weeks. Items are answered on a 5-point Likert-scale from 0 'not at all' to 4 'extremely'. Total scores range from 0 to 28, with higher scores reflective of greater insomnia severity. Scores of 8 or greater indicate the presence of at least mild clinical insomnia.
Executive function | Pre-intervention
  Executive function will be measured with the Trail Making Test (TMT), a paper-and-pencil neuropsychological instrument comprised of two parts, A and B. Time taken to complete each part is calculated in seconds, with longer times indicative of poorer performance. To minimize practice effects, comparable alternative forms will be used for post-intervention assessments.
Memory | Pre-intervention
  Memory will be measured with the Verbal Paired Associates I and II (VPAI and VPAII) tasks, subtests included in the Wechsler Memory Scale - Fourth Edition (WMS-IV) neuropsychological battery. VPAI assesses immediate recall of verbally-presented associated word pairs and VPAII measures delayed, long-term memory. Performance is evaluated by comparing the number of correctly recalled word pairs with age-based norms, with higher scores indicative of better verbal memory.
Attention and psychomotor performance | Pre-intervention
  Attention and psychomotor performance will be measured with the Coding task, a subtest included in the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV). Participants use a key to match as many numbers to corresponding nonsense symbols as possible within a two-minute time limit. Performance is evaluated by comparing the total number of correct matches to age-based norms, with higher scores indicative of better attention and psychomotor functioning.
Decision making assessed by the IGT | Pre-intervention
  Decision making will be measured with three self-administered computerized tasks. The Iowa Gambling Task (IGT) produces a score representative of risky decision making by assessing participants' tendency to choose more disadvantageous over advantageous selections. For this measure, lower scores represent greater risky decision making.
Decision making assessed by the MCQ | Pre-intervention
  Decision making will be measured with three self-administered computerized tasks. The Monetary Choice Questionnaire (MCQ) is a measure of delay-discounting designed to assess preferences for smaller, more immediate rewards over larger, delayed rewards. An average score is produced based on participant responses to 27 trials, with higher values indicative of steeper discounting of delayed rewards and greater impulsivity.
Decision making assessed by the GDT | Pre-intervention
  Decision making will be measured with three self-administered computerized tasks. The Game of Dice Task (GDT) produces a score representative of risky decision making by assessing participants' tendency to choose more disadvantageous over advantageous selections. For this measure, lower scores represent greater risky decision making.
Anxiety | Change from pre-intervention to 2 weeks post-intervention
  Anxiety symptoms will be measured with the 14-item self-report Hospital Anxiety and Depression Scale (HADS). This instrument assesses symptoms of anxiety and depression specifically among patients with physical illnesses. Seven items assess symptoms of anxiety, while the remaining 7 items assess symptoms of depression. Each item is scored on a 4-point Likert-scale ranging from 0 to 3. Subscale scores, ranging from 0 to 21, can be calculated for anxiety and for depression, with higher scores indicative of greater symptoms.
Depression | Change from pre-intervention to 2 weeks post-intervention
  Depressive symptoms will be measured with the 14-item self-report Hospital Anxiety and Depression Scale (HADS). This instrument assesses symptoms of anxiety and depression specifically among patients with physical illnesses. Seven items assess symptoms of anxiety, while the remaining 7 items assess symptoms of depression. Each item is scored on a 4-point Likert-scale ranging from 0 to 3. Subscale scores, ranging from 0 to 21, can be calculated for anxiety and for depression, with higher scores indicative of greater symptoms.
HF-related quality of life | Change from pre-intervention to 2 weeks post-intervention
  HF-related quality of life will be measured with the 23-item self-report Kansas City Cardiomyopathy Questionnaire (KCCQ), a HF-specific measure designed to quantify physical limitations, symptoms, and HF-related quality of life. The measure includes 9 subscales that can be combined into an overall summary score ranging from 0-100, with higher scores indicative of better functioning and fewer symptoms.
HF self-care | Change from pre-intervention to 2 weeks post-intervention
  HF self-care will be measured with the 15-item self-report Self Care of Heart Failure Index (SCHFI). This instrument assesses patient's adherence to specific HF dietary and symptom monitoring guidelines, their confidence in adhering to these guidelines, and the steps they take when they notice changes in their symptom status. Three subscales (Management, Maintenance, and Confidence) are scored out of 100, with higher scores representing better self-care.
Executive function | Change from pre-intervention to 2 weeks post-intervention
  Executive function will be measured with the Trail Making Test (TMT), a paper-and-pencil neuropsychological instrument comprised of two parts, A and B. Time taken to complete each part is calculated in seconds, with longer times indicative of poorer performance. To minimize practice effects, comparable alternative forms will be used for post-intervention assessments.
Memory | Change from pre-intervention to 2 weeks post-intervention
  Memory will be measured with the Verbal Paired Associates I and II (VPAI and VPAII) tasks, subtests included in the Wechsler Memory Scale - Fourth Edition (WMS-IV) neuropsychological battery. VPAI assesses immediate recall of verbally-presented associated word pairs and VPAII measures delayed, long-term memory. Performance is evaluated by comparing the number of correctly recalled word pairs with age-based norms, with higher scores indicative of better verbal memory.
Attention and psychomotor performance | Change from pre-intervention to 2 weeks post-intervention
  Attention and psychomotor performance will be measured with the Coding task, a subtest included in the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV). Participants use a key to match as many numbers to corresponding nonsense symbols as possible within a two-minute time limit. Performance is evaluated by comparing the total number of correct matches to age-based norms, with higher scores indicative of better attention and psychomotor functioning.
Decision making assessed by the MCQ | Change from pre-intervention to 2 weeks post-intervention
  Decision making will be measured with three self-administered computerized tasks. The Monetary Choice Questionnaire (MCQ) is a measure of delay-discounting designed to assess preferences for smaller, more immediate rewards over larger, delayed rewards. An average score is produced based on participant responses to 27 trials, with higher values indicative of steeper discounting of delayed rewards and greater impulsivity.
Decision making assessed by the GDT | Change from pre-intervention to 2 weeks post-intervention
  Decision making will be measured with three self-administered computerized tasks. The Game of Dice Task (GDT) produces a score representative of risky decision making by assessing participants' tendency to choose more disadvantageous over advantageous selections. For this measure, lower scores represent greater risky decision making.
Functional Status | Change from pre-intervention to 2 weeks post-intervention
  Functional status will be measured with the Sixty-Foot Walk Test (60ftWT), an ambulatory measure that requires patients to walk four laps of 15 feet. Time needed to walk each of the four laps, as well as the total duration, is recorded in seconds, with higher completion times indicative of poorer functional status.
Insomnia severity | Change from pre-intervention to 6 months post-intervention
  Insomnia symptoms will be measured with the 7-item self-report Insomnia Severity Index (ISI). This measure assesses the severity of sleep-onset and sleep maintenance difficulties, sleep satisfaction, as well as associated daytime dysfunction and distress over the prior two weeks. Items are answered on a 5-point Likert-scale from 0 'not at all' to 4 'extremely'. Total scores range from 0 to 28, with higher scores reflective of greater insomnia severity. Scores of 8 or greater indicate the presence of at least mild clinical insomnia.
Sleep quality assessed by the PSQI | Change from pre-intervention to 6 months post-intervention
  Sleep quality will be measured with the 19-item self-report Pittsburgh Sleep Quality Index (PSQI). Seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction) are derived from the instrument which can then be summed to produce a total 'global' PSQI score ranging from 0 to 21. Total PSQI scores greater than 5 indicate poor sleep quality.
Sleep efficiency | Change from pre-intervention to 6 months post-intervention
  Sleep efficiency (SE) will be measured with two-week sleep diaries where participants log their daily bed and wake times, as well as the number of hours of sleep each night. SE will be calculated as the percentage of sleep time divided by time spent in bed, with higher percentages indicative of more efficient sleep.
Anxiety | Change from pre-intervention to 6 months post-intervention
  Anxiety symptoms will be measured with the 14-item self-report Hospital Anxiety and Depression Scale (HADS). This instrument assesses symptoms of anxiety and depression specifically among patients with physical illnesses. Seven items assess symptoms of anxiety, while the remaining 7 items assess symptoms of depression. Each item is scored on a 4-point Likert-scale ranging from 0 to 3. Subscale scores, ranging from 0 to 21, can be calculated for anxiety and for depression, with higher scores indicative of greater symptoms.
Depression | Change from pre-intervention to 6 months post-intervention
  Depressive symptoms will be measured with the 14-item self-report Hospital Anxiety and Depression Scale (HADS). This instrument assesses symptoms of anxiety and depression specifically among patients with physical illnesses. Seven items assess symptoms of anxiety, while the remaining 7 items assess symptoms of depression. Each item is scored on a 4-point Likert-scale ranging from 0 to 3. Subscale scores, ranging from 0 to 21, can be calculated for anxiety and for depression, with higher scores indicative of greater symptoms.
HF-related quality of life | Change from pre-intervention to 6 months post-intervention
  HF-related quality of life will be measured with the 23-item self-report Kansas City Cardiomyopathy Questionnaire (KCCQ), a HF-specific measure designed to quantify physical limitations, symptoms, and HF-related quality of life. The measure includes 9 subscales that can be combined into an overall summary score ranging from 0-100, with higher scores indicative of better functioning and fewer symptoms.
HF self-care | Change from pre-intervention to 6 months post-intervention
  HF self-care will be measured with the 15-item self-report Self Care of Heart Failure Index (SCHFI). This instrument assesses patient's adherence to specific HF dietary and symptom monitoring guidelines, their confidence in adhering to these guidelines, and the steps they take when they notice changes in their symptom status. Three subscales (Management, Maintenance, and Confidence) are scored out of 100, with higher scores representing better self-care.
Executive function | Change from pre-intervention to 6 months post-intervention
  Executive function will be measured with the Trail Making Test (TMT), a paper-and-pencil neuropsychological instrument comprised of two parts, A and B. Time taken to complete each part is calculated in seconds, with longer times indicative of poorer performance. To minimize practice effects, comparable alternative forms will be used for post-intervention assessments.
Attention and psychomotor performance | Change from pre-intervention to 6 months post-intervention
  Attention and psychomotor performance will be measured with the Coding task, a subtest included in the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV). Participants use a key to match as many numbers to corresponding nonsense symbols as possible within a two-minute time limit. Performance is evaluated by comparing the total number of correct matches to age-based norms, with higher scores indicative of better attention and psychomotor functioning.
Memory | Change from pre-intervention to 6 months post-intervention
  Memory will be measured with the Verbal Paired Associates I and II (VPAI and VPAII) tasks, subtests included in the Wechsler Memory Scale - Fourth Edition (WMS-IV) neuropsychological battery. VPAI assesses immediate recall of verbally-presented associated word pairs and VPAII measures delayed, long-term memory. Performance is evaluated by comparing the number of correctly recalled word pairs with age-based norms, with higher scores indicative of better verbal memory.
Decision making assessed by the MCQ | Change from pre-intervention to 6 months post-intervention
  Decision making will be measured with three self-administered computerized tasks. The Monetary Choice Questionnaire (MCQ) is a measure of delay-discounting designed to assess preferences for smaller, more immediate rewards over larger, delayed rewards. An average score is produced based on participant responses to 27 trials, with higher values indicative of steeper discounting of delayed rewards and greater impulsivity.
Decision making assessed by the GDT | Change from pre-intervention to 6 months post-intervention
  Decision making will be measured with three self-administered computerized tasks. The Game of Dice Task (GDT) produces a score representative of risky decision making by assessing participants' tendency to choose more disadvantageous over advantageous selections. For this measure, lower scores represent greater risky decision making.
Functional Status | Change from pre-intervention to 6 months post-intervention
  Functional status will be measured with the Sixty-Foot Walk Test (60ftWT), an ambulatory measure that requires patients to walk four laps of 15 feet. Time needed to walk each of the four laps, as well as the total duration, is recorded in seconds, with higher completion times indicative of poorer functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Emery, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No